CLINICAL TRIAL: NCT05529875
Title: Comparison of Propofol and Sevoflurane Anesthesia on the Quality of Recovery After Ambulatory Surgery for Anal Fistula in Obese Patients: A Prospective, Randomized, Single-blinded, Controlled Clinical Trial
Brief Title: Comparison of Propofol and Sevoflurane Anesthesia on the Quality of Recovery After Ambulatory Surgery in Obese Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: In the early stage of the research, this research was limited by the application permission of research drugs and instruments, and the research will have to be interrupted, which is extremely regrettable.
Sponsor: Jiangang Song (Other)
Responsible Party: Sponsor-Investigator, Jiangang Song, Head of Anesthesiology, ShuGuang Hospital
Organization: ShuGuang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20160401
Record Dates: First submitted 2022-05-07; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Quality of Recovery
Keywords: propofol; sevoflurane; obese; quality of recovery; anal fistula
MeSH Terms: conditions — Obesity; Rectal Fistula | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PRO (Active Comparator): Anesthesia was induced by sufentanil citrate 0.2ug/kg and propofol in TCI effect compartment concentration 4-6ug/kg.
  Anesthesia was maintained with propofol in TCI effect compartment concentration 3-4ug/kg.
  Interventions: Drug: Propofol
- Group SEVO (Active Comparator): Anesthesia was induced by sufentanil citrate 0.2ug/kg and sevoflurane in the method of vital capacity with inspired-limb drug concentration measured upon 6%.
  Anesthesia was then maintained with sevoflurane in vaporizer concentration 1.5-2%.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: Propofol — intravenous propofol using target-controlled infusion (TCI) devices.
  Other Names: Group PRO
  Arms: Group PRO
Drug: sevoflurane — inhalator sevoflurane using sevoflurane vaporizer sevoflurane vaporizer.
  Other Names: Group SEVO
  Arms: Group SEVO

SUMMARY:
This study was designed to compare propofol intravenous anesthesia to sevoflurane inhalation anesthesia on the quality of recovery after surgery for anal fistula in obese patients. Propofol-based total intravenous anesthesia (TIVA) and sevoflurane inhalation anesthesia are the two main anesthesia techniques. Obesity influences not only anesthetics metabolic but also physical function of patients, so it is meaningful to study which anesthesia technique is better for the recovery of obese patients after surgery.

DETAILED DESCRIPTION:
This study was approved by Ethical Committee of ShuGuang Hospital affiliated to Shanghai University of Traditional Chinese Medicine. Patients were given informed consent before enrolling the study, whereafter, they were randomized into two groups, propofol-based total intravenous anesthesia (Group PRO) and sevoflurane inhalation anesthesia (Group SEVO). After entering the routine, blood pressure, pulse oxygen saturation, and ECG were monitored by multifunctional anesthesia monitor and anesthesia depth was monitored by brain electrical bispectral index (BIS). Intravenous access (20-gauge catheter) was established and an infusion of lactated Ringer's solution began in the operating room. Patients were positioned as left or right lateral decubitus position according to surgery. Patients inhaled oxygen before anesthetic induction using a face mask. Intravenous penehyclidine hydrochloride 0.5mg, granisetron 3mg, and midazolam 2mg were given as premedication.

In Group PRO, anesthesia was induced by sufentanil citrate 0.2ug/kg and propofol in TCI effect compartment concentration 4-6ug/kg, until the patient loses consciousness, then laryngeal mask airway was inserted. Anesthesia was then maintained with propofol in TCI 3-4ug/kg, if the patient showed body movement, TCI was raised by 0.5 ug/kg every time, until the anesthesia depth was satisfied (no body movement, BIS40-60).

In Group SEVO, anesthesia was induced by sufentanil citrate 0.2ug/kg and sevoflurane. Firstly, mask was fixed with four head band, keeping it sealed. The method of vital capacity was used, taking deep breaths until the patient loses consciousness (call patients not to answer, the eyelash reflex disappeared, BIS40-60): close valve of APL to zero, empty the breathing bag, block the respiratory circuit, prime the circuit with 8% sevoflurane in O2 at 8 L/min until the inspired-limb drug concentration measured upon 6%. Then, laryngeal mask airway was inserted. Anesthesia was then maintained with sevoflurane, adjusting the oxygen flow rate to 2L/min and sevoflurane vaporizer concentration 1.5-2%, if the patient showed body movement and other narcotic lighter sign, sevoflurane vaporizer concentration was raised by 0.5% every time, until the anesthesia depth was satisfied (no body movement, BIS40-60).

The propofol and sevoflurane were closed at the end of surgery.

Quality of recovery was assessed using QoR-40 scale in day 1 and day 2 after surgery. Postoperative pain intensity was assessed using visual analogue scale in day 1 and day 2 after surgery. Surgical and waking time was recorded before leaving post-anesthesia care unit. Adverse events (circulation or respiratory depression, postoperative nausea and vomiting, recovery agitation) were recorded perioperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing selective surgery for anal fistula,
2. aged 18-60 years,
3. body mass index >30kg/m2,
4. patient who required general anesthesia and signed informed consent,
5. ASA I - II.

Exclusion Criteria:

1. patients refused to participate in the test,
2. patients with severe cardiac, pulmonary, liver and renal dysfunction,
3. patients with severe central nervous system diseases or severe mental diseases,
4. patients with a history of alcoholism,
5. allergy to related anesthetics,
6. pregnant or lactating women,
7. participated in the other trials in the past month,
8. taking any sedative, opioid, or sleep aid drugs,
9. patients with other special conditions not suitable for this study, ____________________________________________.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
QoR-40 scales 24 hours after surgery | 24 hours after surgery
  We evaluate the quality of recovery with QoR-40 questionnaire 24 hours after surgery. The Quality of Recovery-40 (QoR-40) questionnaire involves 5 dimensions: physical comfort, physical independence, emotional state, psychological support and pain.
  Dimensions of the QoR-40 identified to represent aspects of good quality recovery after anesthesia and surgery. Positive items were scored from 1(worst) to 5(best); scores were reversed for negative items.
QoR-40 scales 48 hours after surgery | 48 hours after surgery
  We evaluate the quality of recovery with QoR-40 questionnaire 48 hours after surgery. The Quality of Recovery-40 (QoR-40) questionnaire involves 5 dimensions: physical comfort, physical independence, emotional state, psychological support and pain.
  Dimensions of the QoR-40 identified to represent aspects of good quality recovery after anesthesia and surgery. Positive items were scored from 1(worst) to 5(best); scores were reversed for negative items.

SECONDARY OUTCOMES:
Duration of induction | Procedure (After inserting the laryngeal mask airway(LMA ))
  From beginning of intravenous or inhalation of anesthetics to ending of inserting the LMA.
Duration of surgery | Intraoperative
  From beginning of skin cutting to ending of surgery.
Duration of emergence | procedure (After emergence from anesthesia)
  From withdrawl time of intravenous or inhalation of anesthetics to awaking.
visual analogue scales for pain | 1 day (at the time of leaving PACU)
  visual analogue scales for pain in PACU
PONV | 24 hours after surgery
  Postoperative nausea and vomiting in 24hours after surgery
total dosage of Analgesic drugs | 24 hours after surgery
  Categories of analgesics and total dosage of analgesics in 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montgomery JS, Gayed BA, Hollenbeck BK, Daignault S, Sanda MG, Montie JE, Wei JT. Obesity adversely affects health related quality of life before and after radical retropubic prostatectomy. J Urol. 2006 Jul;176(1):257-61; discussion 261-2. doi: 10.1016/S0022-5347(06)00504-0. PMID 16753415
- [Background] Casati A, Putzu M. Anesthesia in the obese patient: pharmacokinetic considerations. J Clin Anesth. 2005 Mar;17(2):134-45. doi: 10.1016/j.jclinane.2004.01.009. PMID 15809132
- [Background] Nakazawa K, Hikawa Y, Maeda M, Tanaka N, Ishikawa S, Makita K, Amaha K. Laryngeal mask airway insertion using propofol without muscle relaxants: a comparative study of pretreatment with midazolam or fentanyl. Eur J Anaesthesiol. 1999 Aug;16(8):550-5. doi: 10.1046/j.1365-2346.1999.00540.x. PMID 10500946
- [Background] Philip BK, Lombard LL, Roaf ER, Drager LR, Calalang I, Philip JH. Comparison of vital capacity induction with sevoflurane to intravenous induction with propofol for adult ambulatory anesthesia. Anesth Analg. 1999 Sep;89(3):623-7. doi: 10.1097/00000539-199909000-00014. PMID 10475291
- [Result] Leger M, Campfort M, Cayla C, Lasocki S, Rineau E. Postoperative quality of recovery measurements as endpoints in comparative anaesthesia studies: a systematic review. Br J Anaesth. 2021 Jun;126(6):e210-e212. doi: 10.1016/j.bja.2021.03.008. Epub 2021 Apr 21. No abstract available. PMID 33892949
- [Result] Niu Z, Gao X, Shi Z, Liu T, Wang M, Guo L, Qi D. Effect of total intravenous anesthesia or inhalation anesthesia on postoperative quality of recovery in patients undergoing total laparoscopic hysterectomy: A randomized controlled trial. J Clin Anesth. 2021 Oct;73:110374. doi: 10.1016/j.jclinane.2021.110374. Epub 2021 Jun 2. PMID 34090183
- [Result] Shen Y, Liu Y, Wu Y, He J. Changes of recovery quality and early cognitive function after treatment of sevoflurane combined with propofol in the elderly undergoing cholecystectomy. Am J Transl Res. 2021 Oct 15;13(10):11868-11874. eCollection 2021. PMID 34786116
- [Result] Senoner T, Velik-Salchner C, Luckner G, Tauber H. Anesthesia-Induced Oxidative Stress: Are There Differences between Intravenous and Inhaled Anesthetics? Oxid Med Cell Longev. 2021 Nov 27;2021:8782387. doi: 10.1155/2021/8782387. eCollection 2021. PMID 34873432
- [Result] Goertz L, Stavrinou P, Hamisch C, Perrech M, Czybulka DM, Mehdiani K, Timmer M, Goldbrunner R, Krischek B. Impact of Obesity on Complication Rates, Clinical Outcomes, and Quality of Life after Minimally Invasive Transforaminal Lumbar Interbody Fusion. J Neurol Surg A Cent Eur Neurosurg. 2021 Mar;82(2):147-153. doi: 10.1055/s-0040-1718758. Epub 2020 Dec 22. PMID 33352610
- [Result] Xu S, Chen JY, Lo NN, Chia SL, Tay DKJ, Pang HN, Hao Y, Yeo SJ. The influence of obesity on functional outcome and quality of life after total knee arthroplasty: a ten-year follow-up study. Bone Joint J. 2018 May 1;100-B(5):579-583. doi: 10.1302/0301-620X.100B5.BJJ-2017-1263.R1. PMID 29701098
- [Result] Zhang Y, Shan GJ, Zhang YX, Cao SJ, Zhu SN, Li HJ, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Propofol compared with sevoflurane general anaesthesia is associated with decreased delayed neurocognitive recovery in older adults. Br J Anaesth. 2018 Sep;121(3):595-604. doi: 10.1016/j.bja.2018.05.059. Epub 2018 Jul 27. PMID 30115258
- [Result] Siampalioti A, Karavias D, Zotou A, Kalfarentzos F, Filos K. Anesthesia management for the super obese: is sevoflurane superior to propofol as a sole anesthetic agent? A double-blind randomized controlled trial. Eur Rev Med Pharmacol Sci. 2015 Jul;19(13):2493-500. PMID 26214787
- [Result] Schwandner O. Obesity is a negative predictor of success after surgery for complex anal fistula. BMC Gastroenterol. 2011 May 23;11:61. doi: 10.1186/1471-230X-11-61. PMID 21605391
- [Result] Cortinez LI, Gambus P, Troconiz IF, Echevarria G, Munoz HR. Obesity does not influence the onset and offset of sevoflurane effect as measured by the hysteresis between sevoflurane concentration and bispectral index. Anesth Analg. 2011 Jul;113(1):70-6. doi: 10.1213/ANE.0b013e31821f105c. Epub 2011 May 19. PMID 21596877
- [Result] Peduto VA, Mezzetti D, Properzi M, Giorgini C. Sevoflurane provides better recovery than propofol plus fentanyl in anaesthesia for day-care surgery. Eur J Anaesthesiol. 2000 Feb;17(2):138-43. doi: 10.1046/j.1365-2346.2000.00626.x. PMID 10758459